CLINICAL TRIAL: NCT07385131
Title: Should Routine Prophylactic Dexamethasone Be Administered Before Intravenous Infliximab in Moderate-to-Severe Inflammatory Bowel Disease: A Prospective, Multicenter, Observational Cohort Study
Brief Title: Prophylactic Dexamethasone Before Infliximab in Moderate-to-Severe IBD
Acronym: PA
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other); First Affiliated Hospital of Wenzhou Medical University (Other); West China Hospital (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); Huzhou Central Hospital (Other); Taizhou Enze Medical Center Group (Other); Lishui Country People's Hospital (Other); Jinhua People's Hospital (Other); Ningbo Medical Center Lihuili Hospital (Other Government); Affiliated Wenling Hospital of Wenzhou Medical University (Other); People's Hospital of Quzhou (Other); Taizhou Municipal Center for Disease Control and Prevention (Unknown); Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0744
Record Dates: First submitted 2026-01-27; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Inflammatory Bowel Disease (IBD); CD - Crohn's Disease; UC - Ulcerative Colitis
Keywords: Infliximab; Dexamethasone; Preventive medication; Infusion reaction
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Dexamethasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- TEST: If there was no allergic reaction during the previous infusion of infliximab, no anti-allergic medication needs to be used before the next infusion.
- DEX: Before each infusion of infliximab, 5mg of dexamethasone was administered intravenously.
  Interventions: Drug: Dexamethasone (IV)

INTERVENTIONS:
Drug: Dexamethasone (IV) — Before each infusion of infliximab, 5mg of dexamethasone was administered intravenously or an equal volume of normal saline was injected.
  Groups: DEX

SUMMARY:
This comparative observational cohort clinical study aims to investigate the necessity of premedication for allergy prevention prior to infliximab injection, and is designed to evaluate whether non-routine administration of dexamethasone before intravenous infusion of infliximab yields greater benefits than routine prophylactic medication in patients with moderate-to-severe inflammatory bowel disease (IBD). This study is designed to optimize the prophylactic strategy prior to Infliximab treatment and advocate for risk stratification-based individualized prophylaxis regimens to avoid hormonal abuse. Additionally, it will construct a risk score using biomarkers to accurately identify high-risk populations in need of prophylaxis and establish a corresponding predictive model. The study is also intended to reduce the use of unnecessary medications, shorten infusion duration and alleviate the medical burden. It is expected to provide targeted clinical support during the early stage of the disease or the course of treatment, improve the efficacy and precision of individualized treatment for patients, and reduce the physical, psychological and economic burdens caused by ineffective treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 14 to 80 years.
* Confirmed cases of inflammatory bowel disease (IBD) with a definitive diagnosis of Crohn's disease (CD) or ulcerative colitis (UC), based on the diagnostic criteria specified in the Chinese Guidelines for the Diagnosis and Treatment of Crohn's Disease (Guangzhou, 2023) and the Chinese Guidelines for the Diagnosis and Treatment of Ulcerative Colitis (Xi'an, 2023). The diagnosis shall be made by comprehensive analysis of clinical manifestations, laboratory tests, imaging examinations, endoscopic examinations and histopathological findings, with infectious colitis and other non-infectious colitis ruled out.
* Moderate to severe CD: for adults aged 18 years and above, baseline Crohn's Disease Activity Index (CDAI) score >220 or Harvey-Bradshaw Index (HBI) score ≥5; for adolescents aged 14 to 17 years, baseline Pediatric Crohn's Disease Activity Index (PCDAI) score ≥31. Or moderate to severe UC: for adults aged 18 years and above, baseline Mayo score ≥6; for adolescents aged 14 to 17 years, baseline Pediatric Ulcerative Colitis Activity Index (PUCAI) score ≥36.
* Not receiving immunosuppressant therapy (e.g., azathioprine) at present, with no plan to add such medications within the next two months.
* Current glucocorticoid dosage ≤ 10 tablets, and a definite plan has been made for tapering down the dosage to complete discontinuation within the next two months.
* Planned to receive the first dose of infliximab within the next two weeks.

Exclusion Criteria:

* Patients with severe disease who, as judged by the attending clinician, require biological agent intensification therapy, switch therapy or elective surgery within 2 months, such as those with obvious stenosis, perforation, fistula and other conditions leading to obstruction, hemorrhage, infection, etc.
* Patients at high risk of infusion reactions, including those with a history of any biological agent-related infusion reactions, or a history of allergy to any drugs such as penicillins, cephalosporins, sulfonamides, non-steroidal anti-inflammatory drugs (NSAIDs), contrast media, etc.
* Patients with a definite history of food allergy, as well as a past history of asthma or urticaria.
* Patients on chronic daily use of antihistamine antiallergic drugs such as loratadine, cetirizine, diphenhydramine, chlorpheniramine maleate tablets, terfenadine, etc.
* Patients with relative contraindications to biological agents, such as active tuberculosis with positive chest X-ray, strongly positive purified protein derivative (PPD) skin test or positive T-SPOT test; a history of myocardial infarction, heart failure or demyelinating neurological diseases in the past 5 years, etc.
* Patients with relative contraindications to glucocorticoids, such as active tuberculosis, severe infection, gastrointestinal ulcer, etc.
* Patients currently suffering from solid tumors, with a past history of lymphoma or melanoma, or undergoing chemotherapy or radiotherapy.
* Patients complicated with massive gastrointestinal hemorrhage, severe hepatic and renal dysfunction, active bacterial or viral infection, shock, intractable vomiting, severe malabsorption syndrome, etc.
* Patients with psychiatric disorders or insufficient educational level to fully understand the study content.
* Pregnant or lactating patients.
* Patients with severe hemodynamic and vital sign instability, or those with rapidly progressive or end-stage diseases.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with moderate to severe inflammatory bowel disease who are scheduled to receive infliximab treatment for the first time within 2 weeks
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients experiencing infusion reactions | up to the fourth administration of infliximab
  The rate of patients experiencing acute moderate-to-severe infusion reactions related to infliximab during the first four administrations

SECONDARY OUTCOMES:
Concentration of drug and antibody | the 4th and 6th administrations of infliximab
  The changes in the drug concentration and antibody concentration of infliximab during the 4th and 6th administrations, as well as their correlation with the occurrence of infusion reactions.
Severe infusion reactions | through study completion
  The incidence of severe infusion reactions related to infliximab during the first 6 administrations
Hormone-related side effects | through study completion
  The incidence of hormone-related side effects, including hormone-related infections and changes in glycated hemoglobin that occurred throughout the entire study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China